CLINICAL TRIAL: NCT00603993
Title: A Non-Randomized, Open-Label, Roll-Over Study With Self Injection of Adalimumab in Adult Japanese Subjects With Rheumatoid Arthritis
Brief Title: Self-injection of Adalimumab in Adult Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Collaborators: Abbott Japan Co.,Ltd (Industry); Eisai Co., Ltd. (Industry)
Responsible Party: Eiichi Makino, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M05-775
Record Dates: First submitted 2008-01-10; First posted 2008-01-29 (Estimated); Results first posted 2010-02-04 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab (Experimental): Adalimumab 40 mg or 80 mg (same dose subject was receiving in preceding Study M03-651 [NCT 00235872]) subcutaneously (sc) administered every other week (eow) until approval of adalimumab in Japan
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — 40 mg or 80 mg every other week (eow), subcutaneous (sc), self-injection
  Other Names: Humira; ABT-D2E7

SUMMARY:
The purpose of this study is to evaluate the long-term safety of subcutaneous (SC) self-injections (by the subject or subject's family member) of adalimumab in adult Japanese subjects with Rheumatoid Arthritis in an open-label study.

ELIGIBILITY:
Inclusion Criteria:

* Completed Week 36 of Study M03-651 [NCT 00235872]
* Wish to participate in self-injection study
* Give written informed consent
* Comply with protocol requirements

Exclusion Criteria:

* Subject develops serious adverse events at time of eligibility confirmation
* Subject develops severe infections requiring hospitalization or IV injection of antibiotics within 28 days before eligibility confirmation
* Subject develops infections requiring oral administration of antibiotics within 14 days before eligibility confirmation
* The investigator considers the subject inappropriate for participation

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shigeki Hashimoto, PhD, Study Director — Abbott Japan
Locations (16):
- Japan (16):
  - Aichi
  - Chiba
  - Fukuoka
  - Gunma
  - Hokkaido
  - Hyōgo
  - Ibaraki
  - Kanagawa
  - Miyagi
  - Nagano
  - Okayama
  - Osaka
  - Saitama
  - Shizuoka
  - Tokyo
  - Toyama

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab 40 mg or 80 mg Every Other Week (Eow): Adalimumab 40 mg or 80 mg (same dose subject was receiving in preceding Study M03-651 [NCT00235872]) subcutaneously (sc) eow until approval of adalimumab in Japan
Period: Overall Study
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Started | 88
Completed | 68
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
Age Continuous [Mean (Standard Deviation); unit: years] | 52.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 21
Region of Enrollment [Number; unit: participants]
  Japan | 88

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With American College of Rheumatology (ACR) Criteria Improvement of at Least 20%, 50%, and 70% (ACR20/50/70 Responders, Respectively)
Description: Number of responders with ACR criteria improvement consisting of 20%, 50%, and 70% (ACR20, ACR50, and ACR70, respectively) reduction in tender or swollen joint counts (TJC or SJC, respectively) and 20%, 50%, and 70% improvement, respectively, in 3 of the following 5 criteria: [1] physician's global assessment of disease activity (PGA), [2] subject's assessment of disease activity, [3] subject's assessment of pain, [4] subject's assessment of physical disability via a health assessment questionnaire disability index(HAQ-DI), and [5] C-reactive protein (CRP) at each visit.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (Final value)
Population: Analysis was based on observed data.
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
participants
  Week 0 ACR20 | 66
  Week 0 ACR50 | 48
  Week 0 ACR70 | 28
  Week 4 ACR20 | 64
  Week 4 ACR50 | 44
  Week 4 ACR70 | 27
  Week 8 ACR20 | 69
  Week 8 ACR50 | 45
  Week 8 ACR70 | 32
  Week 12 ACR20 | 68
  Week 12 ACR50 | 50
  Week 12 ACR70 | 30
  Week 16 ACR20 | 67
  Week 16 ACR50 | 49
  Week 16 ACR70 | 30
  Week 20 ACR20 | 68
  Week 20 ACR50 | 49
  Week 20 ACR70 | 31
  Week 24 ACR20 | 63
  Week 24 ACR50 | 48
  Week 24 ACR70 | 29
  Week 36 ACR20 | 64
  Week 36 ACR50 | 45
  Week 36 ACR70 | 32
  Week 48 ACR20 | 62
  Week 48 ACR50 | 46
  Week 48 ACR70 | 27
  Week 60 ACR20 | 56
  Week 60 ACR50 | 44
  Week 60 ACR70 | 28
  Week 72 ACR20 | 57
  Week 72 ACR50 | 47
  Week 72 ACR70 | 32
  Week 84 ACR20 | 57
  Week 84 ACR50 | 42
  Week 84 ACR70 | 29
  Week 96 ACR20 | 56
  Week 96 ACR50 | 43
  Week 96 ACR70 | 27
  Week 108 ACR20 | 54
  Week 108 ACR50 | 45
  Week 108 ACR70 | 29
  Week 120 ACR20 | 28
  Week 120 ACR50 | 24
  Week 120 ACR70 | 16
  Week 132 ACR20 | 7
  Week 132 ACR50 | 3
  Week 132 ACR70 | 3
  Final Value ACR20 | 62
  Final Value ACR50 | 49
  Final Value ACR70 | 35

2. Secondary Outcome: Mean Change From Baseline in Tender Joint Count (TJC; Max = 68), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in TJC (max = 68), a component of the ACR criteria, by visit
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (Final value)
Measure: Mean (Standard Deviation); unit: TJC
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
TJC
  Baseline | 20.5 (12.1)
  Week 0 | -15.3 (11.3)
  Week 4 | -14.9 (11.4)
  Week 8 | -15.3 (11.1)
  Week 12 | -14.8 (10.7)
  Week 16 | -14.7 (10.8)
  Week 20 | -15.2 (10.6)
  Week 24 | -15.5 (10.9)
  Week 36 | -14.9 (10.9)
  Week 48 | -15.0 (11.5)
  Week 60 | -15.4 (11.4)
  Week 72 | -15.7 (11.5)
  Week 84 | -16.1 (11.3)
  Week 96 | -16.8 (11.8)
  Week 108 | -16.5 (11.6)
  Week 120 | -18.1 (12.4)
  Week 132 | -19.4 (9.5)
  Final | -14.9 (12.1)

3. Secondary Outcome: Mean Change From Baseline in Swollen Joint Count (SJC, Max = 66), a Component of the ACR Criteria by Visit
Description: Mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in SJC (max = 66), a component of the ACR criteria, by visit
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: SJC
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
SJC
  Baseline | 15.8 (8.6)
  Week 0 | -11.9 (8.3)
  Week 4 | -11.9 (8.3)
  Week 8 | -12.3 (8.0)
  Week 12 | -11.9 (7.7)
  Week 16 | -12.1 (7.8)
  Week 20 | -11.9 (8.3)
  Week 24 | -11.9 (8.3)
  Week 36 | -11.6 (8.3)
  Week 48 | -11.5 (8.8)
  Week 60 | -11.5 (8.4)
  Week 72 | -12.2 (7.8)
  Week 84 | -12.3 (7.8)
  Week 96 | -12.0 (7.8)
  Week 108 | -12.0 (8.2)
  Week 120 | -12.5 (8.7)
  Week 132 | -12.9 (8.0)
  Final | -11.6 (8.0)

4. Secondary Outcome: Mean Change From Baseline in Physician's Global Assessment of Disease Activity (PGA) Using a Visual Analog Scale (0 - 100 mm With 100 mm Being the Worst Assessment), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in PGA (a visual analog scale from 0 - 100 mm with 100 mm being the worst case), a component of the ACR criteria, by visit
Time Frame: Every 4 weeks weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (Final value)
Measure: Mean (Standard Deviation); unit: mm on a scale
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
mm on a scale
  Baseline | 63.2 (21.8)
  Week 0 | -41.0 (26.2)
  Week 4 | -39.5 (27.0)
  Week 8 | -43.3 (23.2)
  Week 12 | -41.6 (24.9)
  Week 16 | -42.1 (25.5)
  Week 20 | -44.0 (24.6)
  Week 24 | -42.3 (26.2)
  Week 36 | -42.2 (25.8)
  Week 48 | -41.4 (27.9)
  Week 60 | -40.7 (28.3)
  Week 72 | -42.2 (26.5)
  Week 84 | -41.9 (26.2)
  Week 96 | -44.6 (24.1)
  Week 108 | -44.7 (25.9)
  Week 120 | -48.8 (27.4)
  Week 132 | -62.4 (10.7)
  Final | -38.8 (31.9)

5. Secondary Outcome: Mean Change From Baseline in Subject's Global Assessment of Disease Activity Using a Visual Analog Scale (0 - 100 mm With 100 mm Being the Worst Assessment), a Component of the ACR Criteria, by Visit
Description: mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in subjects global assessment of disease activity (a visual analog scale from 0 - 100 mm with 100 mm being the worst case), a component of the ACR criteria, by visit
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (Final value)
Measure: Mean (Standard Deviation); unit: mm on a scale
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
mm on a scale
  Baseline | 58.4 (26.8)
  Week 0 | -34.0 (29.8)
  Week 4 | -32.2 (31.1)
  Week 8 | -33.4 (29.2)
  Week 12 | -33.9 (29.3)
  Week 16 | -33.2 (30.9)
  Week 20 | -34.9 (30.4)
  Week 24 | -33.1 (30.9)
  Week 36 | -31.6 (34.6)
  Week 48 | -33.3 (34.0)
  Week 60 | -30.7 (33.6)
  Week 72 | -33.9 (33.1)
  Week 84 | -31.1 (32.2)
  Week 96 | -31.7 (30.4)
  Week 108 | -33.0 (34.0)
  Week 120 | -37.9 (29.4)
  Week 132 | -37.0 (31.7)
  Final | -29.5 (35.7)

6. Secondary Outcome: Mean Change From Baseline in Subject's Assessment of Pain Using a Visual Analog Scale (0 - 100 mm With 100 mm Being the Worst Pain), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in subject's assessment of pain (on a visual analog scale from 0 - 100 mm with 100 mm being the worst pain), a component of the ACR criteria, by visit
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (Final Value)
Measure: Mean (Standard Deviation); unit: mm on a scale
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
mm on a scale
  Baseline | 57.8 (27.1)
  Week 0 | -33.6 (27.7)
  Week 4 | -31.8 (29.6)
  Week 8 | -33.7 (28.1)
  Week 12 | -33.3 (27.7)
  Week 16 | -32.5 (29.7)
  Week 20 | -33.0 (29.9)
  Week 24 | -34.0 (29.3)
  Week 36 | -30.6 (33.3)
  Week 48 | -32.1 (31.7)
  Week 60 | -30.4 (32.8)
  Week 72 | -33.4 (31.2)
  Week 84 | -30.8 (31.3)
  Week 96 | -32.0 (28.3)
  Week 108 | -31.9 (32.1)
  Week 120 | -33.5 (31.1)
  Week 132 | -38.9 (27.1)
  Final | -29.1 (35.8)

7. Secondary Outcome: Mean Change From Baseline in Disability Index of the Health Assessment Questionnaire (HAQ), a Component of the ACR Criteria, by Visit
Description: Mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in disability index of the HAQ (includes 20 questions assessing physical function in 8 domains. The questions are evaluated on a scale from 0 - 3 to measure the ability to perform certain activities [0 = without any difficulty, 1 = with some difficulty, 2 = with much difficulty, and 3 = unable to do so]), a component of the ACR criteria by visit
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (final value)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
units on a scale
  Baseline | 1.4 (0.7)
  Week 0 | -0.5 (0.5)
  Week 4 | -0.5 (0.6)
  Week 8 | -0.6 (0.6)
  Week 12 | -0.6 (0.6)
  Week 16 | -0.6 (0.6)
  Week 20 | -0.6 (0.6)
  Week 24 | -0.6 (0.6)
  Week 36 | -0.5 (0.6)
  Week 48 | -0.6 (0.6)
  Week 60 | -0.5 (0.6)
  Week 72 | -0.6 (0.6)
  Week 84 | -0.5 (0.6)
  Week 96 | -0.5 (0.6)
  Week 108 | -0.6 (0.6)
  Week 120 | -0.6 (0.6)
  Week 132 | -0.7 (0.9)
  Final | -0.5 (0.7)

8. Secondary Outcome: Mean Change From Baseline in C-reactive Protein (CRP), a Component of the ACR Criteria by Visit
Description: Mean change from baseline(for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in CRP (mg/dL), a component of the ACR criteria, by visit
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (Final Value)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 88
mg/dL
  Baseline | 4.0 (2.7)
  Week 0 | -2.5 (2.9)
  Week 4 | -2.4 (3.0)
  Week 8 | -2.5 (2.9)
  Week 12 | -2.6 (2.9)
  Week 16 | -2.6 (2.8)
  Week 20 | -2.8 (2.7)
  Week 24 | -2.8 (2.8)
  Week 36 | -2.8 (3.0)
  Week 48 | -2.7 (3.0)
  Week 60 | -2.3 (3.6)
  Week 72 | -2.5 (3.1)
  Week 84 | -2.7 (3.0)
  Week 96 | -2.8 (2.3)
  Week 108 | -2.9 (2.4)
  Week 120 | -2.8 (2.3)
  Week 132 | -2.9 (1.9)
  Final | -2.2 (4.1)

9. Secondary Outcome: Presence of Morning Stiffness by Visit
Description: The number of subjects with morning stiffness at each visit among those who had morning stiffness at baseline (64).
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (final value)
Population: Subjects were included in this analysis if they had morning stiffness at baseline. Analysis results are as-observed.
Measure: Number; unit: participants
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 64
participants
  Week 0 | 24
  Week 4 | 29
  Week 8 | 26
  Week 12 | 25
  Week 16 | 24
  Week 20 | 23
  Week 24 | 23
  Week 36 | 22
  Week 48 | 19
  Week 60 | 23
  Week 72 | 20
  Week 84 | 21
  Week 96 | 15
  Week 108 | 15
  Week 120 | 7
  Week 132 | 1
  Final | 22

10. Secondary Outcome: Duration (Minutes) of the Presence of Morning Stiffness by Visit
Description: Mean change from baseline (for subjects without rescue treatment, baseline is from Study M02-575 [NCT 00647491]; for subjects with rescue treatment, baseline is from Study M03-651 [NCT 00235872]) in the duration (minutes) of stiffness in the morning.
Time Frame: Every 4 weeks up to Week 24 and every 12 weeks thereafter until study completion or discontinuation (final value)
Population: Subjects were included in this analysis if they had morning stiffness at baseline. Analysis results are as-observed.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Number analyzed (Participants) | 64
minutes
  Baseline | 164.7 (333.9)
  Week 0 | -119.1 (273.0)
  Week 4 | -98.5 (214.8)
  Week 8 | -122.3 (271.8)
  Week 12 | -100.3 (234.9)
  Week 16 | -120.1 (273.3)
  Week 20 | -123.2 (277.2)
  Week 24 | -120.1 (277.8)
  Week 36 | -104.8 (238.0)
  Week 48 | -104.2 (243.7)
  Week 60 | -95.7 (245.8)
  Week 72 | -102.3 (250.4)
  Week 84 | -103.9 (253.4)
  Week 96 | -115.5 (256.2)
  Week 108 | -120.2 (351.8)
  Week 120 | -115.9 (257.3)
  Week 132 | -75.0 (89.8)
  Final | -97.9 (381.3)

ADVERSE EVENTS:
Arm/Group | Adalimumab 40 mg or 80 mg Every Other Week (Eow)
Serious Adverse Events (participants affected / at risk) | 20/88
Other Adverse Events (participants affected / at risk) | 84/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg or 80 mg Every Other Week (Eow) (N=88)
Angina pectoris (Cardiac disorders) | 1
Atrial thrombosis (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Vertigo positional (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Cellulitis (Infections and infestations) | 1
Enteritis infectious (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Ligament rupture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Joint destruction (Musculoskeletal and connective tissue disorders) | 3
Knee deformity (Musculoskeletal and connective tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 4
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab 40 mg or 80 mg Every Other Week (Eow) (N=88)
Anaemia (Blood and lymphatic system disorders) | 7
Vertigo (Ear and labyrinth disorders) | 5
Constipation (Gastrointestinal disorders) | 13
Dental caries (Gastrointestinal disorders) | 11
Diarrhoea (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 6
Gingivitis (Gastrointestinal disorders) | 6
Haemorrhoids (Gastrointestinal disorders) | 6
Stomatitis (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 5
Vomiting (Gastrointestinal disorders) | 5
Adverse drug reaction (General disorders) | 26
Hepatic function abnormal (Hepatobiliary disorders) | 5
Seasonal allergy (Immune system disorders) | 6
Nasopharyngitis (Infections and infestations) | 53
Bronchitis (Infections and infestations) | 12
Upper respiratory tract infection (Infections and infestations) | 9
Pharyngitis (Infections and infestations) | 6
Tinea infection (Infections and infestations) | 5
Contusion (Injury, poisoning and procedural complications) | 11
Fall (Injury, poisoning and procedural complications) | 9
Antinuclear antibody positive (Investigations) | 14
DNA antibody positive (Investigations) | 9
Protein urine present (Investigations) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 5
Headache (Nervous system disorders) | 7
Insomnia (Psychiatric disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 7
Pharyngolaryngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 9
Eczema (Skin and subcutaneous tissue disorders) | 8
Erythema (Skin and subcutaneous tissue disorders) | 5
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 5

LIMITATIONS AND CAVEATS:
Due to the small population, statistical tests were not performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; most restrictive agreement states Medical Institution shall not disclose materials/information disclosed by Abbott Japan in connection with the Clinical Research, or information obtained by conducting the Clinical Research, to third parties without Abbott Japan's prior written approval. When Medical Institution intends to publish information obtained by conducting the Clinical Research, Medical Institution shall obtain Abbott Japan's prior written approval.